CLINICAL TRIAL: NCT00475800
Title: A 39-week, Open-label Extension to CCOX189A2360, a 13-week, Multicenter, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel Trial of 2 Different Dose Regimens of Lumiracoxib (100 mg od and 200 mg od Initial Dose for Two Weeks Followed by 100 mg od) in Patients With Primary Knee Osteoarthritis, Using Celecoxib (200 mg od) as a Comparator
Brief Title: Efficacy and Safety of Lumiracoxib in Patients With Primary Knee Osteoarthritis(OA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCOX189A2360E1
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; lumiracoxib; celecoxib; Cox-2; knee
MeSH Terms: conditions — Osteoarthritis | interventions — lumiracoxib

INTERVENTIONS:
Drug: Lumiracoxib

SUMMARY:
This 39-week, open label study is designed to assess long-term efficacy, safety and tolerability of lumiracoxib 100mg od in patients with osteoarthritis (OA) of the knee who participated in the 13-week core CCOX189A2360 study.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the core CCOX189A2360 study
* Males and females over the 18 years old

Exclusion Criteria:

* Treatment in the extension study is not considered appropriate by the treating physician
* Non-compliance or major protocol violation of the core study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2004-01; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To assess long-term safety and tolerability in patients who were exposed in the core study for 13 weeks to either lumiracoxib, celecoxib or placebo and who will be exposed to lumiracoxib 100 mg od for an additional 39 weeks.

SECONDARY OUTCOMES:
Overall OA pain intensity (Target knee) on a 0-100 mm VAS by visit
Patient's global assessment of disease activity by visit
Physician's global assessment of disease activity by visit.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Tucson, Arizona
  - Brooklyn Park, Minnesota
  - Albuquerque, New Mexico
  - Sioux Falls, South Dakota
  - San Antonio, Texas
- Novartis Investigative Site, Brampton, Ontario, Canada